CLINICAL TRIAL: NCT03736525
Title: DWELL: Design For Wellness - An Online, Randomized Controlled Trial To Create Healthier Home Environments
Brief Title: DWELL: Design For Wellness - An Online Intervention To Create Healthier Home Environments
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laura J. Rosen (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor-Investigator, Laura J. Rosen, Senior Lecturer, Dept. of Health Promotion, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 141.18
Record Dates: First submitted 2018-10-24; First posted 2018-11-09 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Design For Wellness; Wellness
Keywords: Wellness; Home environment; Design; Online intervention; Randomized Controlled Trail (RCT); Nudge theory; Mothers
MeSH Terms: interventions — Research Design; Health

STUDY DESIGN:
Intervention Model Description: Participants will be randomized online to intervention and wait list control groups. Intervention group only will be exposed to a new Facebook group, opened specifically for this study. The Facebook group will have a privacy setting of "closed group", meaning that only members of the group can see posts. This is to prevent possible contamination, ensuring that members of the control group will not be exposed to the intervention. The intervention period will be 3 months. Participants in both groups will fill pre, mid and post intervention questionnaires. At the end of 3 months, we will change the settings of the group and open it to all, including the wait list control group. That way the control group will get access to the treatment as well, to compensate them for participation.
Masking Description: Participants who will be found suitable for participation and who will agree online to participate in the study, will be randomized into intervention and wait list control groups, using an online software "Research Randomizer". The wait list control group will not receive any special treatment during the study. Both groups will be asked to answer the online questionnaires, and after the end of the intervention period the wait list control group will get access to the Facebook group also, to compensate them for participation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Design For Wellness (DWELL) (Experimental): Intervention participants will: 1) consume scientific evidence and practical solutions of how to design the home environment for wellness; 2) be part of a community which encourage participants engagement; 3) be empowered to read and control cues in the environment by developing skills.
  Interventions: Behavioral: Design For Wellness (DWELL)
- Wait list control group (Other): After the close of the study, we will open the Facebook group to all, and wait list control group participants can receive a delayed form of the intervention, which includes: 1) consume scientific evidence and practical solutions of how to design the home environment for wellness; 2) be part of a community which encourage participants engagement; 3) be empowered to read and control cues in the environment by developing skills.
  Interventions: Behavioral: Wait list control group

INTERVENTIONS:
Behavioral: Design For Wellness (DWELL) — Design for wellness is an online Facebook intervention. During 3 months intervention period, participants in the intervention group will be exposed to contents on their newsfeed (posts on Facebook wall), and also be expected and encouraged to create new content themselves. The contents will be interactive and involve different modes of delivery, as audio and video, to reinforce active learning. Participants will be part of DWELL Facebook group community and will be empowered to read and control cues in the environment, by developing skills to enhance their self-efficacy.
  Arms: Design For Wellness (DWELL)
Behavioral: Wait list control group — Wait list control group will get no intervention during the study period. Participants will answer questionnaires pre, mid and post intervention. A delayed form of the intervention will be available to them after the close of the study.
  Arms: Wait list control group

SUMMARY:
Design for wellness (DWELL) is an online Facebook intervention developed to effectively cause participants to design their home environments for wellness. Also, to improve health behaviors (specifically: healthy nutrition, physical activity, smoke free home and hygiene); to improve awareness of the importance of the environment in healthy behaviors; and to improve overall wellness. The research will follow qualitative methods in early stages for a deep understanding of participants' needs and inputs, complimented by a rigorous, quantitative approach using randomized controlled trail (RCT) for program evaluation. Participants are Israeli mothers to children up to 18 years old with Facebook profile, who are often in Israel responsible for household management and raising the family. The program will provide the participants with an accessible and convenient online setting for active and group oriented collaborative learning, in informal personalized environment. Motivating the participants to enhance their engagement in DWELL online community is expected to encourage the participants to design their home environment for wellness and improve their health behaviors and overall wellness.

DETAILED DESCRIPTION:
The primary aim of the study is to assess the effectiveness of the intervention on home design for wellness (DWELL). This will be measured through the use of a validated DWELL questionnaire for actions related to changes in home environment for wellness. Secondary aims are to: 1) assess the effectiveness of the intervention on health behaviors, specifically in: nutrition, physical activity, smoke-free homes and hygiene; 2) improve awareness of the importance of the environment in healthy behavior; 3) improve wellness; 4) assess associations between level of participation (active social, active non-social, passive use) and other outcomes: DWELL, awareness of importance, health behaviors, and wellness.

Participants will be Israeli mothers who are at least 18 years old and have children up to 18 years old, who are willing to participate in the study, can read and write Hebrew, and have internet access and Facebook profile. Recruitment for the trial will be mainly through Facebook and WhatsApp. Semi-structured focus groups will be conducted in order to create DWELL content for intervention and the DWELL questionnaire to assess intervention's effectiveness.

A randomized controlled trial (RCT) will be conducted to assess effectiveness of an online intervention. Recruitment for the trial will be mainly through Facebook and WhatsApp. Sample size will be calculated based on initial results from the focus group's pilot. After recruitment, participants will be randomised into intervention and wait list control groups, using the online software "Research Randomizer". A three-month Facebook intervention will be carried out. Participants in both groups will fill pre, mid and post intervention questionnaires online. After the first 3 months of the intervention, the investigators will open the group to all participants, including those on the wait list control group. This will allow control group participants to access the treatment and to compensate the participants for participation. The investigators will continue to follow and manage the group and monitor its long-term activation.

A general linear model will be used which takes in to account repeated measures. A time-to-event analysis using Cox proportional hazards models will be conducted to examine the length of time for which change persisted.

ELIGIBILITY:
Inclusion Criteria:

Israeli mothers who are at least 18 years old and have children <=18 who are willing to participate in a social media (Facebook) intervention.

Exclusion Criteria:

* Participant is not an Israeli woman.
* Participant is not a mother.
* Participant is under 18 years old.
* Participant does not have at least one child up to 18 years old.
* Participant is not willing to participate in the study.
* Participant can not read and write Hebrew.
* Participant does not have internet access.
* Participant does not have Facebook profile. �

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Israeli mothers
Enrollment: 12 (Estimated)
Dates: Start 2018-11-25 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change in home environment design for wellness, as assessed by DWELL questionnaire | Baseline, 6 weeks and 3 months
  DWELL

SECONDARY OUTCOMES:
Change in awareness of the importance of the environment in healthy behaviors, as assessed by DWELL questionnaire | Baseline, 6 weeks and 3 months
  Awareness of the importance of the environment
Changes in Health behaviors, as assessed by existing online questionnaires | Baseline, 6 weeks and 3 months
  Health behaviors: healthy nutrition
Changes in Health behaviors, as assessed by existing online questionnaires | Baseline, 6 weeks and 3 months
  Health behaviors: physical activity
Changes in Health behaviors, as assessed by existing online questionnaires | Baseline, 6 weeks and 3 months
  Health behaviors: smoke-free homes
Changes in Health behaviors, as assessed by existing online questionnaires | Baseline, 6 weeks and 3 months
  Health behaviors: good hygiene
Change in overall wellness, as assessed by WHO-5 instrument | Baseline, 6 weeks and 3 months
  Overall wellness
Change in overall wellness, as assessed by I COPPE instrument | Baseline, 6 weeks and 3 months
  Overall wellness
level of participation in the online Facebook group (active social, active non-social, passive use) will be associated with the outcome: DWELL | Baseline, 6 weeks and 3 months
  Level of participation
level of participation in the online Facebook group (active social, active non-social, passive use) will be associated with the outcome: awareness of importance of design for wellness | Baseline, 6 weeks and 3 months
  Level of participation
level of participation in the online Facebook group (active social, active non-social, passive use) will be associated with the outcome: health behaviors | Baseline, 6 weeks and 3 months
  Level of participation
level of participation in the online Facebook group (active social, active non-social, passive use) will be associated with the outcome: wellness | Baseline, 6 weeks and 3 months
  Level of participation

CONTACTS AND LOCATIONS:
Overall Officials: Tal Aperman-Itzhak, PhD Student, Study Director — School of Public Health, Dept. of Health Promotion, Sackler Faculty of Medicine, Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Ramat Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aperman-Itzhak T, Prilleltensky I, Rosen L. Improving Knowledge, Engagement, and Self-Efficacy in the Creation of Healthy Home Environments for Mothers Using a Facebook Intervention (Design for Wellness): Randomized Controlled Trial. J Med Internet Res. 2023 Nov 7;25:e46640. doi: 10.2196/46640. PMID 37934566